CLINICAL TRIAL: NCT05993767
Title: Pharmacokinetic Study of an Optimized Dose Ratio of Dolutegravir/Emtricitabine/Tenofovir Alafenamide Fumarate: Expediting a UNIVERSAL First Line Regimen for All Children Living With HIV in Africa
Brief Title: UNIVERSAL 1: Pharmacokinetic Study of a Novel DTG/FTC/TAF Dose Ratio for Children
Acronym: UNIVERSAL1
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PENTA Foundation (Network)
Collaborators: Radboud University Medical Center (Other); Baylor College of Medicine (Other); Clinton Health Access Initiative Inc. (Other); University of Zimbabwe (Other); Chiang Mai University (Other); Joint Clinical Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNIVERSAL1; RIA2019PD-2882 (Other Grant/Funding Number: EDCTP2)
Record Dates: First submitted 2023-08-01; First posted 2023-08-15 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; Clinical Protocols; Emtricitabine

STUDY DESIGN:
Intervention Model Description: An interventional, phase I/II, multicenter, single-arm study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- dolutegravir (DTG)/emtricitabine (FTC)/tenofovir alafenamide (TAF) regimen (Experimental): Switch or start dolutegravir (DTG)/emtricitabine (FTC)/tenofovir alafenamide (TAF) regimen with a novel dose ratio for HIV treatment. Subjects will receive DTG 10 mg dispersible tablets and FTC/TAF 15/1.88 mg dispersible tablets or DTG 50 mg film coated tablets and FTC/TAF 200/25 mg film coated tablets depending on weight band
  Interventions: Drug: dolutegravir (DTG)/emtricitabine (FTC)/tenofovir alafenamide (TAF) regimen; Drug: Dolutegravir (DTG)/ Emtricitabine (FTC)/tenofovir alafenamide (TAF)

INTERVENTIONS:
Drug: dolutegravir (DTG)/emtricitabine (FTC)/tenofovir alafenamide (TAF) regimen — Switch or start dolutegravir (DTG)/emtricitabine (FTC)/tenofovir alafenamide (TAF) regimen with a novel dose ratio for HIV treatment
Drug: Dolutegravir (DTG)/ Emtricitabine (FTC)/tenofovir alafenamide (TAF) — Single arm

SUMMARY:
This study aims to find out whether treating children living with HIV with three anti-HIV medicines, dolutegravir (DTG), emtricitabine (FTC) and tenofovir alafenamide (TAF), with a novel dose ratio will achieve adequate drug concentrations and is safe. The optimal DTG/FTC/TAF dose ratio will be used for the development of a fixed-dose combination dispersible tablet.

DETAILED DESCRIPTION:
Dolutegravir (DTG), Emtricitabine (FTC) and Tenofovir alafenamide (TAF) are anti-HIV medicines. DTG works very well, can be taken once-daily and has few side effects. In international treatment guidelines, DTG is one of the most recommended medicines for adults and young people. Emtricitabine is also one of the preferred medicines in anti-HIV treatment for adults and children. Tenofovir alafenamide (TAF) is not yet recommended in children <25 kg, however TAF could potentially be used safely and effectively in children.

Combining DTG, FTC and TAF in a specific dose ratio may offer treatment that is safe and effective. If so, a combination dispersible tablet containing these three medicines can be developed and this will allow the same HIV medicines to be used across children and adults.

This study will include 50 children aged 28 days to less than 10 years old who are living with HIV. All participants will receive the same treatment with DTG, FTC and TAF. Subjects will receive DTG 10 mg dispersible tablets and FTC/TAF 15/1.88 mg dispersible tablets or DTG 50 mg film coated tablets and FTC/TAF 200/25 mg film coated tablets depending on weight band. All children in the study will have clinical assessments. Blood tests will be performed to make sure that the medicines are safe and, at some visits, participants and carers will also be asked to answer some questions on taking medicine and how medicine tastes. All children will be followed up for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 28 days and 10 years old
* Weighing 3 to <25 kg
* Confirmed HIV-1 infection (local, molecular methods)
* A parent or legal guardian is willing and able to give informed consent on behalf of the child as per national legislation and willing to adhere to the protocol
* Participant is willing to give informed assent if the trial site clinician deems them old enough and able to understand the age-appropriate information about participation in the study
* Girls who have reached menarche must have a negative pregnancy test at screening
* Subject is willing to start DTG/FTC/TAF regimen in the novel dose ratio for HIV treatment
* Subjects already on a DTG-based ART regimen should be virologically suppressed at screening

Exclusion Criteria:

* Age between 28 days and 10 years old
* Weighing 3 to <25 kg
* Confirmed HIV-1 infection (local, molecular methods)
* A parent or legal guardian is willing and able to give informed consent on behalf of the child as per national legislation and willing to adhere to the protocol
* Participant is willing to give informed assent if the trial site clinician deems them old enough and able to understand the age-appropriate information about participation in the study
* Girls who have reached menarche must have a negative pregnancy test at screening
* Subject is willing to start DTG/FTC/TAF regimen in the novel dose ratio for HIV treatment
* Subjects already on a DTG-based ART regimen should be virologically suppressed at screening
* History or presence of known allergy to DTG, FTC or TAF
* Alanine aminotransferase (ALT) ≥5 times the upper limit of normal (ULN), OR ALT ≥3xULN AND bilirubin ≥2xULN
* Patients with severe hepatic impairment or unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice), known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Current or anticipated need for TB therapy during the study
* Use of rifampicin-based therapy within 4 weeks before start trial
* Presence of comedication known to interact with trial medications
* Known resistance to INSTI or NRTI

Ages: 28 Days to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary endpoints for DTG: | From enrollment to the end of treatment at 24 weeks
  - Geometric mean Ctrough concentration
Primary endpoints for DTG: | From enrollment to the end of treatment at 24 weeks
  Percentage of individual Ctrough concentrations below the 90% effective concentration (EC90) (0.32 mg/L)
Primary endpoints for DTG: | From enrollment to the end of treatment at 24 weeks
  - Geometric mean DTG Ctrough, Cmax, and AUC
Primary safety endpoints | From enrollment to the end of treatment at 24 weeks
  - Occurrence of serious adverse events
Primary safety endpoints | From enrollment to the end of treatment at 24 weeks
  - Occurrence of new clinical and laboratory grade 3 and 4 adverse events
Primary safety endpoints | From enrollment to the end of treatment at 24 weeks
  Occurrence of adverse events (of any grade) leading to treatment modification
Primary endpoints for FTC/TAF: | From enrollment to the end of treatment at 24 weeks
  - Geometric mean Ctrough, Cmax, and AUC
Primary endpoints for FTC/TAF: | From enrollment to the end of treatment at 24 weeks
  Intracellular tenofovir diphosphate (TDP) levels at 24 hours acquired through dried blood spot analysis

SECONDARY OUTCOMES:
Efficacy endpoints | From enrollment to the end of treatment at 24 weeks
  - Viral load (VL) <400 c/ml at 24 weeks
Efficacy endpoints | From enrollment to the end of treatment at 24 weeks
  Occurrence of new or recurrent WHO clinical stage 3 or 4 event

CONTACTS AND LOCATIONS:
Locations (3):
- Uganda (2):
  - Baylor College of Medicine Children's Foundation, Kampala
  - Joint Research Centre, Kampala
- University of Zimbabwe Clinical Research Centre, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No
IPD will be supporting a generic company dossier subject to FDA evaluation